CLINICAL TRIAL: NCT06282276
Title: Anti-fat Attitudes and Weight Stigma Among Orthopedic Surgeons and Their Correlation to the Therapeutic Approach to Patients With Obesity
Brief Title: Anti-fat Attitudes and Weight Stigma Among Orthopedic Surgeons
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 012922HYMC
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Weight Stigma
MeSH Terms: conditions — Weight Prejudice | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: cross sectional survey — filling out the electronic survey form

SUMMARY:
Evidence shows that anti-fat attitudes and weight stigma are prevalent among healthcare professionals and may affect treatment decisions regarding patients with obesity. The present study aimed to examine the presence of anti-fat attitudes and weight stigma among orthopedic surgeons and their correlation to the therapeutic approach to patients with obesity. In this cross-sectional survey, 150 orthopedic surgeons will complete a web-based questionnaire. the questionnaire is based on Antifat Attitudes Questionnaire (AFA), developed by Crandall in 1994. In addition, the questionnaire will include a questionnaire developed by Bocquier in 200521 to explore weight stigma among physicians.

DETAILED DESCRIPTION:
Data will be collected through an online questionnaire consisting of four parts. Part 1 will gather socio-demographic data using nine items. Part 2 will utilize the Antifat Attitudes Questionnaire (AFA), developed by Crandall in 1994. The questionnaire, comprising 13 items, will assess three subscales:1. "Dislike" measuring explicit antipathy toward fat individuals.2. "Fear of Fat" measuring personal concerns about weight or becoming overweight.3. "Willpower" measuring beliefs about personal control over being overweight. Participants will rate items on a 10-point Likert scale, with higher scores indicating greater anti-fat bias. Part 3 will include a questionnaire developed by Bocquier in 2005 to explore weight stigma among physicians, consisting of 12 items. Participants will rate items on a 6-point Likert scale, with higher scores indicating stronger weight stigma. Part 4 will investigate the therapeutic approach of orthopedic surgeons to patients with obesity using five items. Participants will items on a 6-point Likert scale, with higher scores indicating a stronger preference for a conservative approach.

ELIGIBILITY:
Inclusion Criteria: orthopedic surgeon age 18 till 80 -

Exclusion Criteria:

-

Ages: 25 Years to 72 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 150 orthopedic surgeon's
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
anti fat attitudes | 3 months
  Orthopedic surgeons' personal beliefs about weight
Weight stigma | 3 months
  Orthopedic surgeons' personal beliefs about weight
Therapeutic approach | 3 months
  Orthopedic surgeons' magnitude of preference for a conservative approach when treating patients with obesity

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Research data may be available on a reasonable request